CLINICAL TRIAL: NCT02416921
Title: Preventing Weight Gain in African American Reproductive-Aged Women: Pilot Program
Brief Title: Preventing Weight Gain in African American Reproductive-Aged Women
Acronym: FB--Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Missouri, Kansas City (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201412141; 1P30DK092950 (NIH)
Record Dates: First submitted 2015-03-18; First posted 2015-04-15 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Weight Gain; Women's Health; Obesity
Keywords: Facebook; Weight Gain Prevention; Women's Health; Online; Weight Gain; Weight Loss; Female Contraception; Obesity; Body Weight; Internet
MeSH Terms: conditions — Weight Gain; Obesity; Weight Loss; Body Weight | interventions — Women's Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weight-gain Prevention (Experimental): Subjects in this group will engage in a 4-week weight-gain prevention curriculum delivered via Facebook
  Interventions: Behavioral: Weight-gain Prevention
- Women's Health (Active Comparator): Subjects in this group will engage in a 4-week women's health curriculum delivered via Facebook
  Interventions: Behavioral: Women's Health

INTERVENTIONS:
Behavioral: Weight-gain Prevention — A 4-week weight-gain prevention curriculum will be delivered via Facebook. Participants will be provided tips to prevent weight-gain and will be given the opportunity to engage with the peer coaches and other participants in the group.
  Arms: Weight-gain Prevention
Behavioral: Women's Health — A 4-week women's health curriculum will be delivered via Facebook. Participants will be provided tips for staying healthy and will be given the opportunity to engage with the peer coaches and other participants in the group.
  Arms: Women's Health

SUMMARY:
The purpose of this research study is to evaluate the effect of a Facebook-delivered weight-gain prevention program versus a Facebook-delivered program with general women's health information.

DETAILED DESCRIPTION:
Weight gain is an important health concern, and disparities in the prevalence of obesity between African American and White women increase throughout the reproductive period. This study is a randomized, controlled trial testing the feasibility and acceptability of a peer-coach-administered, Facebook-delivered intervention to prevent weight gain in overweight and obese African American women. Study visits lasting approximately 1 hour will occur at baseline, post-intervention, and 1-month follow-up, to assess effectiveness and acceptability. The core intervention will occur over a 4-week period. Educational content in both the weight-gain prevention program and women's health program will be delivered via Facebook, with new content posted each weekday related to that week's topics. The peer coaches may contact participants via private messaging, when needed, to provide support and encourage engagement. If successful, this intervention could be easily disseminated to populations in under-served and community settings.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Has Facebook account and uses it, on average, at least once a day
* Body Mass Index (BMI) of 25-45
* Has access to the internet
* Able to consent in English

Exclusion Criteria:

* Currently pregnant or breastfeeding, recently postpartum (within 6 weeks)
* Diagnosis of Diabetes Mellitus
* History of contraindicated medical conditions or conditions that can affect weight
* Current use of certain medications

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Program satisfaction, as measured by the OWN Program Satisfaction Survey | 9 weeks, beginning with start of cohort

CONTACTS AND LOCATIONS:
Overall Officials: Rick Stein, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States